CLINICAL TRIAL: NCT00038116
Title: Embryonic Dopamine Cell Implants for Parkinson's Disease: A Double-Blind Study
Brief Title: Embryonic Dopamine Cell Implants for Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 93-0097
Record Dates: First submitted 2002-05-29; First posted 2002-05-30 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; PD; dopamine; embryonic dopamine cell implant surgery; tissue implants
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- embryonic dopamine cell implant surgery (Active Comparator): embryonic dopamine cell implant surgery
  Interventions: Procedure: embryonic dopamine cell implant surgery
- sham surgery (Placebo Comparator): sham surgery (placebo)
  Interventions: Procedure: placebo

INTERVENTIONS:
Procedure: embryonic dopamine cell implant surgery — Half of the participants received the cell implant surgery, while the other half received the placebo. After the double-blind phase of the study, patients in the placebo group had the option of receiving tissue implants. Fourteen of these patients eventually had transplants.
  Arms: embryonic dopamine cell implant surgery
Procedure: placebo — sham surgery
  Arms: sham surgery

SUMMARY:
The purpose of this trial is to determine if patients who received embryonic dopamine cell implant surgery showed significantly greater improvement in their Parkinson's disease than a control group undergoing the placebo treatment, and to determine if the cell implant surgery was more effective in younger or older patients.

DETAILED DESCRIPTION:
Parkinson's disease is caused by the death of a small number of nerve cells that produce a critical chemical called dopamine. The drug L-dopa can partially make up for the lack of dopamine. As time goes on, however, most patients notice that the drugs do not work as well. Oftentimes, patients develop great fluctuations in motor control. Off drugs they cannot move, and on drugs they have excess, exaggerated movements. Research in animals over the last 20 years has shown that dopamine cells can be replaced by transplants of new cells obtained from fetal brain tissue. For the past 14 years, several laboratories around the world have been performing similar transplants of human fetal brain tissue on patients with Parkinson's disease. So far, it has been impossible to compare results from the different groups because no two centers are performing transplants in the same way.

This study seeks to get around that problem using a controlled clinical trial that compares the embryonic dopamine cell implant surgery with a placebo treatment. A total of 40 patients were recruited--half received the cell implant surgery, while the other half received the placebo. After the double-blind phase of the study, patients in the placebo group had the option of receiving tissue implants. Fourteen of these patients eventually had transplants. At present, this study is providing long-term follow-up evaluation and treatment for the subjects.

ELIGIBILITY:
INCLUSION CRITERIA:

* Idiopathic Parkinson's disease of at least 7 years duration and responsive to levodopa. Other Parkinson syndromes excluded.
* Patients previously tried on other available forms of medical treatment.
* Age between 20 and 75 years.
* Presence of an intractable problem, such as "off" periods, dyskinesias, or "freezing," not controlled by dopamine agonists such as levodopa or pergolide.
* No serious depression and no cognitive impairment.
* Successful completion of home diary by patient or responsible party.
* Successful videotape recordings at home of "on" and "off" status.
* Normal MRI of brain within the last 18 months.
* Fluorodopa PET scan compatible with idiopathic Parkinson's disease.
* Medically fit to undergo implant surgery with certification by the patient's physician.
* Able to financially cover expenses not paid for by NIH grant (between $1,000 and $2,000 for unreimbursed travel, video camera, and blood screening as specified in the consent form.

EXCLUSION CRITERIA:

* Severe or moderately severe depression or cognitive impairment.
* Previous brain surgery.
* Presence of diabetes mellitus, severe cardiopulmonary disease or other severe medical disease, or MRI evidence of cerebrovascular disease.
* Not medically cleared to undergo a surgical procedure.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1995-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
a subjective Global Rating Scale | duration of the trial

SECONDARY OUTCOMES:
objective measurements of PD, including UPDRS motor "off", Schwab and England "off", and 19F-fluorodopa uptake | duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Curt R. Freed, M.D., Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University Hospital, the University of Colorado Health Sciences Center, Denver, Colorado
  - North Shore University Hospital, Manhasset, New York
  - The Movement Disorder Center, Columbia-Presbyterian Hospital, New York, New York

REFERENCES:
- [Background] Freed CR, Greene PE, Breeze RE, Tsai WY, DuMouchel W, Kao R, Dillon S, Winfield H, Culver S, Trojanowski JQ, Eidelberg D, Fahn S. Transplantation of embryonic dopamine neurons for severe Parkinson's disease. N Engl J Med. 2001 Mar 8;344(10):710-9. doi: 10.1056/NEJM200103083441002. PMID 11236774
- [Background] Nakamura T, Dhawan V, Chaly T, Fukuda M, Ma Y, Breeze R, Greene P, Fahn S, Freed C, Eidelberg D. Blinded positron emission tomography study of dopamine cell implantation for Parkinson's disease. Ann Neurol. 2001 Aug;50(2):181-7. doi: 10.1002/ana.1075. PMID 11506400
- [Background] Ma Y, Feigin A, Dhawan V, Fukuda M, Shi Q, Greene P, Breeze R, Fahn S, Freed C, Eidelberg D. Dyskinesia after fetal cell transplantation for parkinsonism: a PET study. Ann Neurol. 2002 Nov;52(5):628-34. doi: 10.1002/ana.10359. PMID 12402261
- [Background] Trott CT, Fahn S, Greene P, Dillon S, Winfield H, Winfield L, Kao R, Eidelberg D, Freed CR, Breeze RE, Stern Y. Cognition following bilateral implants of embryonic dopamine neurons in PD: a double blind study. Neurology. 2003 Jun 24;60(12):1938-43. doi: 10.1212/01.wnl.0000070181.28651.3b. PMID 12821736
- [Background] Bjorklund A, Dunnett SB, Brundin P, Stoessl AJ, Freed CR, Breeze RE, Levivier M, Peschanski M, Studer L, Barker R. Neural transplantation for the treatment of Parkinson's disease. Lancet Neurol. 2003 Jul;2(7):437-45. doi: 10.1016/s1474-4422(03)00442-3. No abstract available. PMID 12849125
- [Background] Freed CR, Leehey MA, Zawada M, Bjugstad K, Thompson L, Breeze RE. Do patients with Parkinson's disease benefit from embryonic dopamine cell transplantation? J Neurol. 2003 Oct;250 Suppl 3:III44-6. doi: 10.1007/s00415-003-1308-5. PMID 14579124
- [Background] Gordon PH, Yu Q, Qualls C, Winfield H, Dillon S, Greene PE, Fahn S, Breeze RE, Freed CR, Pullman SL. Reaction time and movement time after embryonic cell implantation in Parkinson disease. Arch Neurol. 2004 Jun;61(6):858-61. doi: 10.1001/archneur.61.6.858. PMID 15210522
- [Background] McRae C, Cherin E, Yamazaki TG, Diem G, Vo AH, Russell D, Ellgring JH, Fahn S, Greene P, Dillon S, Winfield H, Bjugstad KB, Freed CR. Effects of perceived treatment on quality of life and medical outcomes in a double-blind placebo surgery trial. Arch Gen Psychiatry. 2004 Apr;61(4):412-20. doi: 10.1001/archpsyc.61.4.412. PMID 15066900
- [Result] Ma Y, Tang C, Chaly T, Greene P, Breeze R, Fahn S, Freed C, Dhawan V, Eidelberg D. Dopamine cell implantation in Parkinson's disease: long-term clinical and (18)F-FDOPA PET outcomes. J Nucl Med. 2010 Jan;51(1):7-15. doi: 10.2967/jnumed.109.066811. Epub 2009 Dec 15. PMID 20008998